CLINICAL TRIAL: NCT01128725
Title: Truncated and Extended Forms of Amyloid Beta Peptides in Alzheimer's Disease: Genesis, Toxicity and Identification as Biological Markers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 10-PP-01
Record Dates: First submitted 2010-05-21; First posted 2010-05-24 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2010-05

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Group Alzhamyd (Other): The patients coming in consultation for a mnésique complaint will see each other offering the study. During a consultation, the following balance sheet will be accomplished :clinical Maintenance, collection of records and used treatments
  * psycho-behaviour Valuation through Neuropsychiatric Inventory (NPI) and through Inventory Apathy
  * Valuation of self-government in the activities of daily life (IADL). Further to this balance sheet, it is habitually offered on the subjects of advice (principally centered on the proposals of use of external helps for instance book memo, agenda and internal assistants medium notes-techniques and associations to keep information) and a new consultation 1 year afterwards including the same balance sheet.
  In a supplementary way in this clinical valuation, a blood sample will be accomplished at the time of inclusion and 12 months afterwards.
  Interventions: Other: Alzhamyd

INTERVENTIONS:
Other: Alzhamyd — The patients coming in consultation for a mnésique complaint will see each other offering the study. During a consultation, the following balance sheet will be accomplished :clinical Maintenance, collection of records and used treatments
  * psycho-behaviour Valuation through Neuropsychiatric Inventory (NPI) and through Inventory Apathy
  * Valuation of self-government in the activities of daily life (IADL). Further to this balance sheet, it is habitually offered on the subjects of advice (principally centered on the proposals of use of external helps for instance book memo, agenda and internal assistants medium notes-techniques and associations to keep information) and a new consultation 1 year afterwards including the same balance sheet.
  In a supplementary way in this clinical valuation, a blood sample will be accomplished at the time of inclusion and 12 months afterwards.

SUMMARY:
Beta amyloid immunoreactivity is probably due to a significant number of Ab catabolites corresponding to N-terminally truncated and Cterminally truncated or extended forms which display distinct propensity to aggregation. Very few things are known concerning the mechanisms and proteases by which they are generated. Furthermore, the link between truncation and toxicity has not been delineated.

Finally, little is known concerning Ab fragments in biological fluids and whether they could be seen as early biomarkers and thereby, as putative targets for AD diagnostic. The present project will allow to examine the human biological samples and to identify various cohorts after complete clinical evaluation.

ELIGIBILITY:
Inclusion Criteria:

* 1) Coming subjects to see patients in CMRR for a complaint mnésique 2) Introducing a score in Tiny Mental the upper Test (MMSE) in 28/30 without error in under score of the recall of the 3 words 3) Introducing a score of 10/10 in the test of the 5 words of B2C 4) Introducing a score in the ladder CDR (Clinical Dementia Rating) equal to 0 5) Having given a lit consent 6) Being affiliated member or beneficiary of the regime of French national health and pensions organization

Exclusion Criteria:

* Major, all the vulnerable persons under 18 under tutelage, under legal guardianship, deprived of freedom, hospitalized in a health Establishment or social for quite other reason that searches it
* Record of neurological or psychiatric pathology and inability for sensory reasons to perform a cognitive balance sheet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-09; Primary Completion 2010-09 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Identification of yet unknown enzymes involved in the processing of Ab, especially on those responsible for the exoproteasic truncation of Ab at its N-terminus. | one year
  Identification of yet unknown enzymes involved in the processing of Ab, especially on those responsible for the exoproteasic truncation of Ab at its N-terminus.

SECONDARY OUTCOMES:
The availability of truncated fragments designed to set up monoclonal antibodies will allow us to estimate their associated toxicity in various cellular models. | one year
  Secondly, the availability of truncated fragments designed to set up monoclonal antibodies will allow us to estimate their associated toxicity in various cellular models. Furthermore, we will be able to compare the toxicity of soluble monomers and aggregates. Third, we expect to determine the content of these Ab species in the biological fluids of various representative non-demented or AD affected patients.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe ROBERT, Principal Investigator — CHU de Nice - CM2R - Hôpital de Cimiez - 4 avenue reine victoria - 06 003 Nice cedex 1
Locations (1):
- Robert, Nice, Alpes-Maritimes, France